CLINICAL TRIAL: NCT02327221
Title: A Phase IIb, Multicentre, Randomised, Double-blinded, Placebo-controlled, Multi-dose and Multi-injection, Parallel Groups Study to Evaluate the Efficacy and the Safety of Ovasave in Patients With Active Refractory Crohn's Disease
Brief Title: Study Evaluating Ovasave, an Autologous Cell Therapy, in Patients With Active Crohn's Disease
Acronym: CATS29
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: TxCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXC-CD-002-2011; 2014-001295-65 (EudraCT Number)
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Cell therapy; Regulatory T lymphocytes; Treg; Autologous; Antigen specific T regulatory lymphocytes
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ovasave - Dose 10e4 (Active Comparator)
  Interventions: Drug: Ovasave
- Ovasave - Dose 10e6 (Active Comparator)
  Interventions: Drug: Ovasave
- Ovasave - Dose 10e7 (Active Comparator)
  Interventions: Drug: Ovasave
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ovasave — During CATS29-Double blind phase, two intravenous administrations of study drug will be administered, one at week 0 and another one at week 8.
  Arms: Ovasave - Dose 10e4; Ovasave - Dose 10e6; Ovasave - Dose 10e7
Drug: Placebo — During CATS29-Double blind phase, two intravenous administrations of study drug will be administered, one at week 0 and another one at week 8.
  Arms: Placebo

SUMMARY:
The investigational product, named Ovasave (Ova-Treg), is a cell-based therapy, consisting of an autologous antigen-specific regulatory type 1 T lymphocyte expanded population administered via the intravenous route as an infusion.

The study is a multicenter, randomised, double-blinded, placebo-controlled, multi-dose and multi-injection study; followed with a 16-week phase with either the possibility for an open-label treatment part or a safety follow-up part with no injection.

Then, the patients will be followed in an additional long-term safety follow-up, of maximum duration of 3 years from the first administration.

DETAILED DESCRIPTION:
During double-blinded phase, the treatment consists of 2 intravenous (i.v.) administrations of antigen-specific autologous T regulatory cells or placebo:

* Group A: 1.10e4 cells and 1.10e4 cells
* Group B: 1.10e6 cells and 1.10e6 cells
* Group C: 1.10e7 cells and 1.10e7 cells
* Group D: Placebo and Placebo

During double-blinded phase, two i.v. administrations of study drug (Ova-Treg) will be administered, one at week 0 and another one at week 8 for the group A, B and C. Two injections of Placebo will be administered, one at week 0 (V4) and another one at week 8 for the group D. During double-blinded phase, all the patients will be followed during 16 weeks. This will be followed by an additional period of 16 weeks when the patient is expected to receive two additional administrations of Ovasave at 10e6 cells dose (Open-label phase), except if refused by the patient or not recommended by the Investigator, representing the follow-up phase. These third and fourth administrations will be performed for all groups (A, B, C and D) with an injection of Ovasave at 1.10e6 cells administered at week 16 and week 24. A patient who didn't receive the 2 first administrations during the double-blinded phase cannot receive the third and the fourth administration during Open-label phase.

ELIGIBILITY:
Main Inclusion Criteria:

1. Active Crohn's Disease diagnosis defined as patients with medical history of signs, symptoms and biological evidence of active bowel inflammation:

   * Documented endoscopic evidence of inflammatory bowel disease (IBD), compatible with Crohn's diagnosis at least 1 year prior to screening and
   * High sensitive C-reactive protein (hs-CRP) > 10 mg/L at V1.
2. Failure or intolerance to conventional treatments including corticosteroid, immunosuppressant and at least one biologics; and had not responded (primarily failure) or responded and then lost response completely (no response or need to increase the dose / secondary failure) or were intolerant to this therapy at a dose indicated for CD
3. Documented CDAI (Crohn's Disease Activity Index) above 250 points (CDAI ≥ 250) at screening or within the past 3 months;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
CDAI response | 6 weeks post administration
  Controlled versus placebo confirmation of the ability of a single intravenous (i.v.) injection of 1.10e6 cells dose of Ovasave (Ova-Treg cells) to induce a CDAI response (CDAI decrease ≥ 100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Severine VERMEIRE, MD, Principal Investigator — UZ Gasthuisberg, Gent (Belgium)
Locations (29):
- Austria (2):
  - Medical University Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
  - CHU Liege, Liège
- France (11):
  - CHU d'Amiens Sud, Amiens
  - CHU de Besançon, Hôpital Jean Minjoz, Besançon
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - CHRU de Lille, Hôpital Claude Huriez, Lille
  - CHU de Nancy, Hôpital de Brabois Adulte, Nancy
  - CHU de Nice, Hôpital de l'Archet 2, Nice
  - Hôpital Saint-Louis, Paris
  - Hôpital St-Antoine, Paris
  - CHU de Bordeaux, Hôpital Haut-Lévêque, Pessac
  - CHU de Toulouse, Hôpital Rangueil, Toulouse
- Germany (6):
  - Krankenhaus Waldfriede e.V., Berlin
  - Markus Hospital, Frankfurt am Main
  - Hannover Medical School, Hanover
  - University Hospital Schleswig-Holstein, Kiel
  - Gastroenterologische Gemeinschaftpraxis, Minden
  - Universitätsklinik Ulm, Ulm
- Italy (4):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Clinico Humanitas, Milan
  - Complesso Integrato Columbus, Roma
  - Ospedale San Camillo-Forlanini, Roma
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Background] Desreumaux P, Foussat A, Allez M, Beaugerie L, Hebuterne X, Bouhnik Y, Nachury M, Brun V, Bastian H, Belmonte N, Ticchioni M, Duchange A, Morel-Mandrino P, Neveu V, Clerget-Chossat N, Forte M, Colombel JF. Safety and efficacy of antigen-specific regulatory T-cell therapy for patients with refractory Crohn's disease. Gastroenterology. 2012 Nov;143(5):1207-1217.e2. doi: 10.1053/j.gastro.2012.07.116. Epub 2012 Aug 8. PMID 22885333